CLINICAL TRIAL: NCT03440528
Title: Using of Irradiated Amnion Dressing for the Treatment of Skin Ulcer
Status: Completed | Type: Observational
Sponsor: Egyptian Atomic Energy Authority (Other Government)
Collaborators: Waleed Nemr,Egyptian Atomic Energy Authority (Unknown)
Responsible Party: Principal Investigator, Nashwa Radwan, Lecture of Dermatology, Egyptian Atomic Energy Authority
Other Study IDs: 29112017NCRRT
Record Dates: First submitted 2017-12-30; First posted 2018-02-22 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Ulcer
Keywords: Skin ulcer, Human amniotic membrane, Treatment
MeSH Terms: conditions — Ulcer; Skin Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the using of a commercial product of dried human amniotic membrane sterilized by gamma irradiation for the treatment of skin ulcer.

DETAILED DESCRIPTION:
Dried human amniotic membrane patches were obtained from National center for radiation research and technology, Egypt, under commercial name REGE pro.

ELIGIBILITY:
Inclusion Criteria:

* patients have unhealing ulcer

Exclusion Criteria:

* must stop other line of treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study is based on randomized selection of 3 types of ulcer ( diabetic foot ulcer, post operative ulcer and ultrasonic ulcer)
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Size of ulcer | 2 week
  REGE pro decreased size of ulcer after second treatment

SECONDARY OUTCOMES:
Reduction of pain | 1 week
  Patients response revealed reduction of pain at the time of application. One week post application, a questionnaire were collected from patients; about 95% of them ensured that pain was controlled.

OTHER OUTCOMES:
Complete curring | 4 to 10 weeks
  REGE pro healed ulcer after 4 to 10 weeks. The improvement of ulcer was observed by photographs taken before and each week post application.
Freedom from scarring | 10 weeks
  It was observed that the using of REGE pro prevent any scar formation in all applied patients.

CONTACTS AND LOCATIONS:
Overall Officials: Nashwa K Radwan, PhD, Study Director — NATIONAL CENTER FOR RADIATION RESEARCH AND TECHNOLOGY
Locations (1):
- Amniotic tissue lab, Cairo, Egypt